CLINICAL TRIAL: NCT02348164
Title: Human Lycopene and Beta-cryptoxanthin Absorption From Citrus Fruit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FL62 Citrus Study
Record Dates: First submitted 2015-01-21; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Bioavailability of Carotenoids
Keywords: Carotenoids; absorption; citrus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 (Experimental): Volunteers receive pink grapefruit first followed by tangerines two weeks later
  Interventions: Other: Pink grapefruit first followed by tangerines two weeks later
- Treatment 2 (Experimental): Volunteers receive tangerines first followed by pink grapefruit two weeks later
  Interventions: Other: Tangerines first followed by pink grapefruit two weeks later

INTERVENTIONS:
Other: Pink grapefruit first followed by tangerines two weeks later — A 504 gram serving of pink grapefruit was fed as a single meal followed by 234 grams tangerines two weeks later
  Arms: Treatment 1
Other: Tangerines first followed by pink grapefruit two weeks later — A 234 gram serving of tangerines was fed as a single meal followed by 504 grams pink grapefruit two weeks later
  Arms: Treatment 2

SUMMARY:
The goal of the research study is to measure and compare the absorption of equivalent amounts of beta-cryptoxanthin and Iycopene provided in citrus fruit. The investigators want to determine whether adults absorb beta-cryptoxanthin to a greater extent than lycopene, when both are supplied in comparable citrus fruits.

DETAILED DESCRIPTION:
Lycopene and beta-cryptoxanthin are carotenoids found in a small number of foods. Unlike lycopene, beta-cryptoxanthin is among the 10% of carotenoids that can form vitamin A. Lycopene is primarily found in tomatoes and tomato-based products, but also in pink grapefruit and pink guava. Beta-cryptoxanthin is primarily found in tangerines, oranges, pumpkin, peaches, and papayas. Tomatoes and tomato products contain very high concentrations of lycopene, but beta-cryptoxanthin is present in modest amounts, of about 2 to 3 mg per serving, even in its primary food sources. Lycopene is typically the most abundant carotenoid in the diet and in the blood. Despite its scarcity in foods, beta-cryptoxanthin is the third or fourth most abundant carotenoid in blood.

This suggests that beta-cryptoxanthin absorption and metabolism may be quite different from the absorption and metabolism of lycopene and other carotenoids. Specifically, it suggests either that beta-cryptoxanthin itself is absorbed unusually well or that the citrus fruits that are the primary food sources of beta-cryptoxanthin in the diet are much more bioavailable than the tomato products that are the major source of lycopene. The investigators hypothesize that adults absorb a significantly greater amount of beta-cryptoxanthin than lycopene even when both carotenoids are supplied in comparable amounts in a similar matrix.

Subjects will be given a list of foods that are good sources of lycopene and beta-cryptoxanthin and asked to avoid them. Both carotenoids are found in limited numbers of foods, and can be avoided by limiting intakes of tomatoes, red and orange peppers, pumpkin, watermelon, pink guava, pink grapefruit, tangerines, oranges, papayas and mangos. The investigators will feed citrus fruit to volunteers in a randomized crossover design. On study days 14 and 28, subjects will receive either tangerines, or pink grapefruit in a randomized fashion so that each subject gets both treatments during the study. Each subject will serve as his/her own control, and will be fed both treatments at different times, separated by a two-week washout period.

On days 14 and 28, subjects will arrive at the Western Human Nutrition Research Center at approximately 10:30 AM. After a baseline blood draw, subjects will be fed their carotenoid-containing fruit with a controlled meal (low carotenoid, 30-35% fat). Subjects will be given a controlled, low carotenoid, 30-35% kcal from fat dinner at about 6:30 PM on treatment days (days 14 and 28) and a controlled low carotenoid, 30 - 35% kcals from fat breakfast at about 8 AM on study days 15 and 29. Investigators will collect 25 mL of blood per collection, by venipuncture of an arm vein at the following time points, 0, 3, 5, 7, 9, 21, and 24hr following the fruit containing meal. Blood will be collected into heparinized vacutainer tubes and placed on ice in a covered ice bucket.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Body mass indexes between 18 and 35
* Blood pressure under 150/90 mm Hg
* Not pregnant, lactating, or planning a pregnancy within 90 days.

Exclusion Criteria:

* Total cholesterol concentrations over 250 mg/dL
* Total fasting triacylglycerol concentrations over 175 mg/dL.
* Taking lipid-lowering medications (gemfibrozil, niacin, lovastatin, simvastatin)
* Taking fat blocking medications (such as orlistat)
* Taking medicines containing high dosages of retinoids such as Accutane
* Taking carotenoid dietary supplements
* Known allergy to tangerines or pink grapefruit
* Consuming more than 2 alcoholic drinks per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change in carotenoid appearance in blood following fruit ingestion | Day 14 - 0, 3, 5, 7, 9, 21, and 24hr after meal
  Carotenoids (lycopene, lutein, beta-carotene and beta-cryptoxanthin), vitamin A and vitamin E will be measured with reverse-phase liquid chromatography diode array detection.
Change in carotenoid appearance in blood following fruit ingestion | Day 28 - 0, 3, 5, 7, 9, 21, and 24hr after meal
  Carotenoids (lycopene, lutein, beta-carotene and beta-cryptoxanthin), vitamin A and vitamin E will be measured with reverse-phase liquid chromatography diode array detection.

SECONDARY OUTCOMES:
Change in blood lipids following meal ingestion | Day 14 - 0, 3, 5, 7, 9, 21, and 24hr after meal
  Total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides will be measured with an automated Hitachi analyzer
Change in blood lipids following meal ingestion | Day 28 - 0, 3, 5, 7, 9, 21, and 24hr after meal
  Total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides will be measured with an automated Hitachi analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Betty J Burri, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States